CLINICAL TRIAL: NCT05162716
Title: Cardiac ResynchrOniSation Via Stimulation of the LEFT Bundle in AF Patients.
Acronym: CROSS-LEFT-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nicolas Clementy, MD, PhD (Other)
Collaborators: Dr Arnaud BISSON (Unknown)
Responsible Party: Sponsor-Investigator, Nicolas Clementy, MD, PhD, Associate Professor, University Hospital, Tours
Organization: University Hospital, Tours (Other)
Other Study IDs: CROSS-LEFT AF
Record Dates: First submitted 2021-12-08; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Pacing-Induced Cardiomyopathy
Keywords: left bundle branch area pacing; atrial fibrillation; atrioventricular ablation; pacing-induced cardiomyopathy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LBBAP: Patients with permanent atrial arrhythmia with an indication of cardiac pacing and atrioventricular junction ablation will undergo the implantation of a single-chamber pacemaker with left bundle branch area pacing, and then atrioventricular junction ablation.
  Interventions: Device: Single-chamber pacemaker implantation with left bundle branch area pacing

INTERVENTIONS:
Device: Single-chamber pacemaker implantation with left bundle branch area pacing — A prepectoral single-chamber pacemaker is implanted with a 3830 (Medtronic) IS-1 pacing lead screwed via the right ventricle in the deep interventricular septum in order to capture the left Purkinje system on the left ventricular endocardial side.
  Other Names: Atrioventricular junction ablation

SUMMARY:
Permanent ventricular pacing may be complicated with ventricular dyssynchrony and subsequent pacing-induced cardiomyopathy. We hypothesized that left bundle branch area pacing may prevent the development of pacing-induced cardiomyopathy in patients with permanent atrial fibrillation requiring permanent ventricular pacing.

Patients with permanent atrial arrhythmia with an indication of cardiac pacing and atrioventricular junction ablation will be prospectively enrolled.

They will undergo the implantation of a single-chamber pacemaker with left bundle branch area pacing, and then atrioventricular junction ablation.

They will be prospectively followed during 6 months.

DETAILED DESCRIPTION:
Patients with permanent atrial arrhythmia with an indication of cardiac pacing and atrioventricular junction ablation will be prospectively enrolled.

They will undergo the implantation of a single-chamber pacemaker with left bundle branch area pacing confirmed according to electrocardiographic parameters. Atrioventricular node ablation will be performed the following day through a femoral venous approach.

Perioperative data and potential complications will be collected. Patients will be prospectively followed during 6 months. They will have clinical examination, 12-lead ECG, and an echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Permanent atrial arrhythmia
* Symptoms related to an insufficient rate control under optimal medical therapy

Exclusion Criteria:

* Indication of prophylactic defibrillator
* Already implanted with a cardiac device

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated with pacemaker implantation and atrioventricular junction ablation for symptomatic chronic atrial arrhythmia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Heart failure hospitalization | 6 months
  Hospitalization for decompensated heart failure

SECONDARY OUTCOMES:
Mortality | 6 months
  Death from any cause
Electrical remodeling | 6 months
  QRS width
Complications | 30 days
  Perioperative complications
Volumetric response | 6 months
  Left ventricular ejection fraction, left ventricular volumes

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Tours, Tours, Please Select..., France

IPD SHARING:
Plan to Share IPD: Undecided